CLINICAL TRIAL: NCT00785551
Title: A Single-Dose, Open-Label Comparative Study of the Pharmacokinetics, Safety,and Tolerability of Oral Quinine Sulfate in Healthy Volunteers and Adults With Mild and Moderate Renal Impairment
Brief Title: Comparative Study of Quinine Sulfate in Healthy Patients and in Patients With Renal Impairment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-001-07-1008
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Healthy; Renal Impairment
Keywords: male; female; pharmacokinetics; normal and impaired renal function
MeSH Terms: conditions — Renal Insufficiency | interventions — Quinine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): quinine sulfate 648mg in subjects with normal renal function (CLcr > 80mL/min)
  Interventions: Drug: quinine sulfate
- 2 (Experimental): quinine sulfate 648mg in subjects with mildly impaired renal function (CLcr > 50 to 80 mL/min)
  Interventions: Drug: quinine sulfate
- 3 (Experimental): quinine sulfate 648mg in subjects with moderately impaired renal function (CLcr 30 to 50mL/min)
  Interventions: Drug: quinine sulfate

INTERVENTIONS:
Drug: quinine sulfate — 2 x 324mg given in one dose to healthy subjects
  Other Names: Qualaquin
  Arms: 1
Drug: quinine sulfate — 2 x 324mg given as one dose to subjects with mild renal impairment
  Other Names: Qualaquin
  Arms: 2
Drug: quinine sulfate — 2 x 324mg given as one dose to subjects with moderate renal impairment
  Other Names: Qualaquin
  Arms: 3

SUMMARY:
The effects of mild or moderate renal impairment (creatinine clearance 30 to 50 ml/min or >50 to 80 ml/min, respectively) on the pharmacokinetic profile of quinine and its active metabolite, 3'-hydroxyquinine, will be investigated. Safety and tolerability in healthy subjects versus those with mild to moderate renal impairment will be compared, as well.

DETAILED DESCRIPTION:
Since many of the adverse events associated with quinine are dose-related, it is important to consider how varying degrees of renal dysfunction alter quinine pharmacokinetics possibly warranting dosage adjustment in these patients. This study will compare the pharmacokinetics of quinine in patients with normal, mild or moderate renal impairment. Eighteen non-smoking males and female volunteers between 18-65 years of age weighing at least 60 kg with BMI between 18- 40 kg/m2 will be divided into 3 groups of 6 subjects each based on renal function as defined (6 normal, 6 mild impairment, 6 moderate impairment). Subjects will be confined to the study unit during the entire 5 day study period beginning on the evening of Day -3. To confirm renal function classification, creatinine clearance will be measured via 24-hour urine collection from 7am Day -2 until 7am Day -1. On day 1, after a fast of at least 8 hours, each patient will receive a single 648 mg dose of quinine sulfate. Blood and urine samples will be collected at times sufficient to adequately define the pharmacokinetics of quinine and its active metabolite, 3'-hydroxyquinine) in the three study groups. Subjects will be monitored regarding adverse effects throughout study participation.

ELIGIBILITY:
Inclusion Criteria:

* All subjects - non-smoking, male and female volunteers 18-65 years of age weighing at least 60kg with BMI between 18- 40kg/m2. Females of childbearing potential sexually inactive or using acceptable birth control method for 14 days prior to through 3 days following dosing or postmenopausal with amenorrhea for at least 2 years, adequate venous access
* Healthy subjects - medically healthy based on designated clinical criteria including CLcr>80 ml/min and hemoglobin 11g/dL or greater
* Renally-impaired subjects - medically acceptable based on designated clinical criteria including good glucose control if diabetic, CLcr 30 to 80 ml/min, hemoglobin 10 g/dL or greater, anticipation that medications necessary for treatment of renal disease and/or other coexisting disease will remain stable for 14 days prior to and throughout the study period

Exclusion Criteria:

* Pregnant or lactating; history of presence of significant cardiovascular, pulmonary, hepatic, hematologic, gastrointestinal, endocrine, immunologic, musculoskeletal, dermatologic, neurologic, or psychiatric disease; positive at screening for HIV, HbsAg, or HCV; QTc >440 msec (male) or 450 msec (female) or PR >200 msec, sitting BP < 90/55, sitting radial pulse < 45 bpm at screening or baseline; history of G6PD deficiency, myasthenia gravis, or optic neuritis; hypersensitivity or idiosyncratic reaction to mefloquine or quinidine; recent/ongoing use of drugs or substances known to inhibit or induce CYP P450 enzymes and/or P-glycoprotein or quinine; hx of alcoholism or drug abuse within previous 2 years; donation of blood or plasma within 56 days prior to dosing; receipt of study medication in another clinical trial within 30 days of dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Alterations pharmacokinetic profile of quinine and 3'-hydroxyquinine in plasma (total and free) and urine following a single 648mg dose of quinine sulfate in healthy subjects with normal renal function versus those with mild and moderate renal impairment | 72 hours

SECONDARY OUTCOMES:
Differences in safety and tolerability of quinine sulfate in healthy subjects versus those with mild and moderate renal impairment | up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davis, M.D., Study Chair — Mutual Pharmaceutical
Locations (1):
- Cetero Research, Miami Gardens, Florida, United States